CLINICAL TRIAL: NCT06009562
Title: Management of Symptomatic Uterine Fibroids in Pregnancy by Laparotomic Myomectomy: a Prospective Cohort Study
Acronym: LPTM-UFs-P
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: University of Palermo (Other)
Responsible Party: Principal Investigator, Andrea Etrusco, M.D., University of Palermo
Other Study IDs: LPTM-S-UFs-Pregancy
Record Dates: First submitted 2023-08-19; First posted 2023-08-24 (Actual); Last update posted 2023-08-24 (Actual); Status verified 2023-08

CONDITIONS: Uterine Fibroid; Pregnancy Related
Keywords: Uterine fibroids; Pregnancy; myomectomy; fetal outcomes
MeSH Terms: conditions — Leiomyoma

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 5 Months
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Procedure: Laparotomic myomectomy during pregnancy — Surgical removal of symptomatic uterine fibroids in pregnancy by laparotomic access

SUMMARY:
The frequency of women presenting with a combination of uterine fibroids and pregnancy is in-creasing nowadays. Uterine fibroids in pregnancy are an unfavorable condition in themselves and being reactive to hormonal stimuli, tending to grow, can generate symptoms of different lev-els of severity. Obstetrics and gynecologists are increasingly faced with the problem of clarifying the management tactics of pregnant patients with symptomatic fibroids, who may see their preg-nancy put at risk by these masses.

ELIGIBILITY:
Inclusion Criteria:

* The large and giant size of UFs, which prevent the proper continuation of pregnancy and/or occupy the entire small and large pelvis, as well as invade and/or occupy the abdominal cavity.
* Circulatory disorders, evidenced by necrosis of the UFs.
* Atypical localization of UFs (cervical, isthmic, intraligamentary, etc.), which caused pelvic organ dysfunction (dysuric phenomena, tenesmus, impediment to the act of defecation, pelvic pain).

Exclusion Criteria:

* Refusal of LPTM by the patient.
* Absence of urgent indication for LPTM during pregnancy.

Sex: Female | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Gender Based: Yes
Study Population: pregnant women with symptomatic uterine fibroids (UFs)
Sampling Method: Non-Probability Sample
Enrollment: 28 (Estimated)
Dates: Start 2023-08-19 (Estimated); Primary Completion 2023-08-19 (Estimated); Study Completion 2024-01-01 (Estimated)

PRIMARY OUTCOMES:
continuation of pregnancy | 5 months
  Pregnancy continuation after surgery.

SECONDARY OUTCOMES:
Fetal outcome | 5 months
  Assessed by APGAR 1 and 5 min, birth weight, and fetal conformation.

CONTACTS AND LOCATIONS:
Overall Officials: Andrea Etrusco, M.D., Principal Investigator — University of Palermo; Antonio Simone Laganà, M.D. Ph.D., Study Director — University of Palermo
Locations (1):
- State-Funded Health Care Facility of Moscow Region (GBUZ MO MONIIAG), Moscow, Russia